CLINICAL TRIAL: NCT06204315
Title: Risk Adapted Spinal Cord/Cauda Constraint Relaxation for High-risk Patients With Metastatic Epidural Spinal Cord Compression Undergoing Spine Stereotactic Radiosurgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Brainlab AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0287; NCI-2024-00049 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord; Metastatic Epidural; Spine Stereotactic
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Radiosurgery (Experimental): A non-invasive, non-surgical procedure that precisely delivers radiation to cancer on the spine while avoiding surrounding, healthy tissue.
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — Given by RTx
  Other Names: CDE-SSRS

SUMMARY:
To learn about the safety of a procedure called cord dose escalated spine stereotactic radiosurgery (CDE-SSRS) in patients with MESCC.

DETAILED DESCRIPTION:
Primary Objectives The primary protocol objectives are to establish the safety of CDE-SSRS alone in participants with MESCC. Specifically, we aim to maintain an RM risk no greater than 1%. RM will be defined as non-functional paresis per the McCormick score (i.e., Grade D).

Secondary Objectives Secondary objectives include pain control as measured by the Brief Pain Inventory, quality of life as measured by the EQ-5D, symptom burden as measured by the MDASI-SP, overall survival, toxicity, ambulatory rate and cost-effectiveness. LC will be defined radiographically with serial MRI scans by the study radiologist per SPINO criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 18 years old
2. Radiographically documented spinal metastasis on spine MRI within 4 weeks of registration
3. Proximity of spinal metastasis to spinal cord or cauda equina which precludes achieving a GTV Dmin of at least 14 Gy per the PI
4. All participants must be able to receive single fraction SSRS at the site of interest with 0.01 cc of the spinal cord receiving 14-16 Gy and/or 0.01 cc of the cauda equina receiving 18-20 Gy. The goal of treatment is to select the minimal dose to the organ at risk which will achieve a GTV Dmin of 14 Gy at the treating physician's discretion.
5. Maximum of 3 contiguous vertebral levels involved with metastasis in the spine to be irradiated in a single session
6. All participants must be able to receive a single fraction spine radiosurgery at the designated site of interest to at least a dose of 18 Gy
7. All participants must have a vertebral level site of interest from C1 to S2
8. Signed informed consent
9. Diagnosis of cancer excluding ultra-radiosensitive histologies (see 4.2)
10. Motor strength ≥ 4 out of 5 in extremity or extremities affected by the level of cord compression
11. ECOG ≤ 2

Exclusion Criteria:

1. Participants with ultra-radiosensitive histologies (lymphoma, multiple myeloma/plasmacytoma)
2. Prior history of radiation at the spinal site of interest
3. Inability to lie supine comfortably for ≥ 60 minutes
4. Progressive neurological deficits due to compression
5. Inability of obtain an MRI
6. Inability or refusal to undergo an MR simulation
7. No eligible for single fraction SSRS for any reason
8. Participants who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Amol Ghia, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org